CLINICAL TRIAL: NCT01051843
Title: Orofacial Difficulties During the Maternal Breastfeeding in Rooming-in
Brief Title: Orofacial Difficulties in Rooming-in
Acronym: AMAC
Status: Completed | Type: Observational
Sponsor: Fortaleza University (Other)
Other Study IDs: AMAC
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-08

CONDITIONS: Orofacial Difficulties in Newborns; Maternal Breastfeeding in Newborns; Newborns in Rooming-in
Keywords: Maternal Breastfeeding; Orofacial Difficulties; Rooming-in; Speech and Language Therapy
MeSH Terms: conditions — Communication Disorders

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to identify the orofacial difficulties during the maternal breastfeeding in rooming-in.

DETAILED DESCRIPTION:
Cross-sectional and quantitative study with sample consisted of 28 dyad present in rooming-in of the Assis Chateaubriand School Motherhood during August and December of 2009.

ELIGIBILITY:
Inclusion Criteria:

* mothers of the newborns participating in the study, regardless of the gender, ethnic and/or age.

Exclusion Criteria:

* newborns who presented oropharyngelarynx structural abnormality, impossibility to feed by mouth and/or exposed in bilispot.

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cross-sectional study of 29 dyads in rooming-in. The data collection consisted in the detection of the main orofacial difficulties during the maternal breastfeeding in rooming-in.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)